CLINICAL TRIAL: NCT04262297
Title: Relation Between Ultrasonographic Rectus Femoris Thickness Measurement and Functionality in Unilateral Transtibial Amputated Prosthesis Users
Brief Title: Rectus Femoris Thickness Measurement in Unilateral Transtibial Amputated Prosthesis Users
Status: Completed | Type: Observational
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Kardelen Gencer Atalay, Principal Investigator, Marmara University
Other Study IDs: 09.2018.025
Record Dates: First submitted 2020-02-06; First posted 2020-02-10 (Actual); Last update posted 2020-02-10 (Actual); Status verified 2020-02

CONDITIONS: Amputation, Traumatic
Keywords: Amputees; Quadriceps MuscleMuscle Strength; Muscle Strength
MeSH Terms: conditions — Amputation, Traumatic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (2):
- Prosthesis users: Prosthesis users with transtibial amputation
- Able-bodied Controls: Prosthesis users' age-, sex- and dominancy-matched healthy controls

SUMMARY:
Knee extension strengthening is one of the cornerstones of rehabilitation in prosthesis users with transtibial amputation. It is recommended in terms of increasing functional mobility, preventing the risk of fall and knee osteoarthritis. Therefore, there is a need for objective measurements to evaluate changes in functional strength and walking through the rehabilitation process. Muscle thickness measured by ultrasound was found to be valid and highly correlated with magnetic resonance imaging and dual-energy X-ray absorptiometry measurements and shown to reflect the strength and functional outcomes in various diseases. The first aim of this study is to reveal the rectus femoris muscle thickness alteration in prosthesis users with transtibial amputation compared to able-bodied controls and establish its correlation with functional strength and walking tests. The second aim is to determine intra- and inter-rater reliability and construct validity of the rectus femoris muscle thickness measured by ultrasound in prosthesis users with transtibial amputation.

DETAILED DESCRIPTION:
Bilateral rectus femoris muscle thickness was measured by two independent examiners using an ultrasound. Bilateral knee extension strength was measured via handheld dynamometer (Jamar, Bolingbrook, IL, USA). Functional strength and walking were assessed by Step-up-over (SUO) and Walk-across (WA) tests of NeuroCom Balance Master® device (NeuroCom International, Clackamas, OR, USA).

ELIGIBILITY:
Inclusion Criteria:

1. Unilateral transtibial amputation on the right side
2. Using the prosthesis for more than 1 year
3. Able to use the prosthesis without pain and discomfort
4. Able to walk without a walking aid

Exclusion Criteria:

1. Presence of concomitant health issues (diabetes mellitus, peripheral artery disease, and other vascular diseases etc.)
2. Ongoing pathology with the contralateral or residual limb (pressure sore or ulcer etc.)
3. Taking medication that is known to affect balance

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Prosthesis users with transtibial amputation and their age-, sex- and dominancy-matched (1:1) able-bodied controls to provide an amputation-independent reference were included.
Sampling Method: Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
Ultrasonographic cross-sectional area of rectus femoris measurement | through study completion, an average of 6 months
  Images were obtained at the bulkiest area of muscle at mid-thigh (midway between the anterior superior iliac spine and the upper pole of the patella) while the participant lay in the supine position with lower limbs are extended and relaxed. The probe was held axially with a light touch in order not to cause any difference in the muscle volume. The rectus femoris cross-sectional area of both limbs (CSA-RF) (mm2) was calculated.

SECONDARY OUTCOMES:
Knee extension strength measurement via handheld dynamometer | through study completion, an average of 6 months
  The dynamometer was located 5 cm above the intermalleolar line to measure bilateral knee extension strength. All participants were tested while lying supine position with a support behind the knees to achieve approximately 30° of flexion. For the amputated-limb, the prosthesis was used in place.
Step-up-over Test | through study completion, an average of 6 months
  All participants were asked to stand still behind the box placed on the pressure platform and to move immediately after seeing the sign on the computer screen. The movement was defined as three phases: first stepping onto the box with one limb, second carrying the body over the box, and third landing with the other limb on the opposite side of the box. The average lift-up index (%), movement time (s), and the impact index for both limbs calculated after three repetitions.
Walk-across Test | through study completion, an average of 6 months
  All participants were asked to stand still and to walk as fast as possible along with the pressure platform after seeing the sign on the computer screen. The average step width (cm), step length (cm), and speed (cm/s) were calculated after three repetitions.

CONTACTS AND LOCATIONS:
Overall Officials: Kardelen Gencer Atalay, Principal Investigator — Marmara University
Locations (1):
- Marmara University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No